CLINICAL TRIAL: NCT07029932
Title: A Randomized, Double-blind, Placebo-controlled, Phase 1 Study of the Safety, Tolerability, and Pharmacokinetics of Single and Multiple Ascending Doses of BWC0977 in Healthy Adult Volunteers
Brief Title: A Phase 1 Study of the Safety and Tolerability of Single and Multiple Ascending Doses of BWC0977 in Healthy Volunteers
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Bugworks Research Inc. (Industry)
Collaborators: Nucleus Network Ltd (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: C003-2025-01; 224842/Z/21/Z (Other Grant/Funding Number: Wellcome Trust); HHS/BARDA OTA No. 75A50122C000 (Other: Biomedical Advanced Research and Development Authority (BARDA)
Record Dates: First submitted 2025-06-12; First posted 2025-06-19 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Infectious Diseases; Antimicrobial Drug Resistance
Keywords: safety; Tolerability; Pharmacokinetics; BWC0977
MeSH Terms: conditions — Communicable Diseases

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, placebo-controlled, combined single and multiple ascending dose (SAD and MAD) trial
Who Masked: Participant, Investigator
Masking Description: Participants will be randomized in a 3:1 ratio of BWC0977 and Placebo. The following controls will be employed to maintain the double-blind status of the study Infusion solution containing active drug and placebo will be indistinguishable in appearance Randomization list will be provided to the study center pharmacist for dispensing purposes and kept in the pharmacy, accessible to the pharmacist and authorized personnel only PK results for the interim analyses between cohorts will be presented in a blinded fashion
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BWC0977 (Experimental): SAD Cohorts: Subjects will receive single doses of BWC0977 via IV infusion over 2 hours. Planned doses to be studied are: 750 mg and 1500 mg.
  MAD Cohorts: Subjects will receive multiple doses of BWC0977 via IV infusion over 30 minutes to 2 hours for 7-10 consecutive days (as per the schedule). Up to four dose groups will be studied. Planned doses and frequencies will be confirmed based on the safety, tolerability, and PK data of BWC0977 obtained in SAD and previous MAD Cohorts
  Interventions: Drug: BWC0977; Drug: Placebo
- Placebo (Placebo Comparator): The placebo used during this study is an active drug formulation without BWC0977.
  SAD Cohorts: Subjects will receive single infusions of placebo in 0.45% sodium chloride for injection over two hours.
  MAD Cohorts: Subjects will receive multiple infusions of placebo in 0.45% sodium chloride for injection over 30 minutes - 2 hours for 7-10 consecutive days (as per schedule). Frequency of infusions will be determined based on safety, tolerability, and PK data obtained for BWC0977 in SAD and previous MAD Cohorts.
  Interventions: Drug: BWC0977; Drug: Placebo

INTERVENTIONS:
Drug: BWC0977 — SAD Cohorts: Double-blind dosing will occur. Six participants will receive single doses of BWC0977. The dose escalation steps may be altered following review of the safety data upon completion of each cohort.
  MAD Cohorts: Double blind dosing will occur. Six participants in each cohort will receive multiple doses of BWC0977. The dose escalation steps may be altered following review of the safety data upon completion of each cohort. Dosing will commence on the morning of Day 1. Dosing frequency to be confirmed based on safety, tolerability, and PK data from SAD and previous MAD cohorts. Daily dosing will continue for a total of 7-10 consecutive days (as per schedule).
Drug: Placebo — SAD Cohorts: Two participants in each cohort will receive a matching placebo. MAD Cohorts: Two participants in each cohort will receive a matching placebo.
  Other Names: active drug formulation without BWC0977

SUMMARY:
The purpose of this study is to assess the safety, tolerability and pharmacokinetics of single and multiple intravenous doses of BWC0977 when administered to healthy adult volunteers.

DETAILED DESCRIPTION:
This Phase 1 study is designed to assess the safety, tolerability, and pharmacokinetics of single and multiple intravenous doses of BWC0977 when administered to healthy adult volunteers. This is a randomized double-blind, placebo-controlled, ascending dose, multi-cohort trial. A total of 64 healthy volunteers are expected to be enrolled in 8 Cohorts. The study will be conducted in two phases: A single ascending dose (SAD) phase, followed by a multiple ascending dose (MAD) phase. In SAD, participants in Cohorts 1 - 2 will receive one dose of BWC0977 or placebo. In MAD, participants in cohorts 3 - 7 will receive multiple doses of BWC0977 or placebo for 7-10 consecutive days (as per the schedule). In both parts, sequential cohorts will be exposed to increasing doses of BWC0977.

ELIGIBILITY:
Inclusion Criteria:

1. Age: Healthy male or female 18 to 55 years of age, inclusive, at time of consent
2. Body mass index (BMI): BMI ≥ 19.0 and ≤ 30.0 (kg/m2) and weight between 55.0 and 100.0 kg (inclusive)
3. Health Status: Medically healthy without significant history of any chronic diseases or conditions (such as cardiovascular, renal, hepatic, neurological, hematological, gastrointestinal, endocrine, or musculoskeletal disorders). Volunteers must have no clinically significant abnormalities in medical history, as determined by the Investigator.
4. Screening Tests:

   1. No findings in Physical examination or vital signs (including temperature, heart rate, respiratory rate, and blood pressure) that the Investigator determines would interfere with interpretation of study results
   2. Triplicate ECGs without clinically significant abnormalities, including a QTcF interval duration ≤450 msec (for males), and ≤470 msec (for females), obtained as an average from the triplicate screening ECGs after at least 5 minutes in a supine, quiet-rest position
   3. For clinically significant abnormalities in the screening clinical laboratory tests, vital signs, and ECG assessments as determined by the Investigator, repeat testing could be performed at the Investigator's discretion
5. Informed consent: Willing and able to provide written informed consent
6. Compliance: Agrees to be available for all study visits and cooperate fully with the requirements of the study protocol, including the schedule of events.
7. Physical Activity Restrictions: Willing to refrain from strenuous physical activity that could cause muscle aches or injury, including contact sports, at any time from 4 days prior to admission in the clinical research unit (CRU) until completion of the study.
8. Venous Access: Have suitable venous access for drug administration and blood sampling
9. Contraception Requirements (for those of reproductive potential): Contraception requirements will follow institutional policies.

   Females:

   Must agree to use two forms of effective contraception-male partner using a condom plus 1 other highly effective method of birth control (e.g., Hormonal methods of contraception including oral contraceptives {includes Combined estrogen-progestin oral contraceptives (COCs) and progestogen-only contraceptives associated with inhibition of ovulation}, a vaginal ring, injectable and implantable hormonal contraceptives, indwelling intrauterine device, history of bilateral tubal ligation, sole vasectomized (bilateral vasectomy) partner with documented azoospermia 90 days after procedure) from signing the consent form until 33 days after last study drug administration, or agree to complete sexual abstinence for the duration of the study from screening and for 33 days after last study drug administration. Females of child-bearing potential must also agree not to donate ova or oocytes (i.e., human eggs) during the study, and for 33 days after completion of the study. For female participants, hormonal contraceptives should begin at least 1 month prior to screening to ensure the contraceptive is in full effect.

   To be considered of non-childbearing potential, a female must have either a hysterectomy, bilateral salpingo-oophorectomy (at least 3 months prior to screening), or menopause {last menstruation >12 months in the absence of other biological causes and follicle-stimulating hormone levels in menopausal range (>40mIU/mL)}, provision of written documentation is not required for female sterilization and oral confirmation is adequate. Female participants in same sex relationships do not need to utilize contraception.

   Males:

   If sexually active with a female partner of childbearing potential, must agree to use male condom plus 1 other highly effective method of birth control in their partner (e.g., Hormonal methods of contraception including oral contraceptives {includes Combined estrogen-progestin oral contraceptives (COCs) and progestogen-only contraceptives associated with inhibition of ovulation}, a vaginal ring, injectable and implantable hormonal contraceptives, indwelling intrauterine device, history of bilateral tubal ligation) from signing the consent form until 93 days after last study drug administration, or agree to complete sexual abstinence for the duration of the study from screening and for 93 days after last study drug administration. Hormonal contraceptives should be in use by female partner for at least 1 month prior to screening to ensure contraceptive is in full effect.

   To be considered surgically sterile, male participants must have had bilateral vasectomy at least 3 months before screening with appropriate documentation of the absence of sperm in the ejaculate 90 days after procedure. The use of condom by male partner will be required if bilateral vasectomy is the chosen highly effective method of birth control.

   Male participants must also agree not to donate sperms during the study and for 93 days after the last dose of the study drug.

   Male participants in same sex relationships or sexually active with female of non-childbearing potential (as defined above) do not need to utilize contraception. Male participants with potentially postmenopausal partners who are under the age of 55 years must use condoms unless their partner's postmenopausal status has been confirmed by FSH level

   Exclusion Criteria:
   * 1) Pregnancy and Lactation: Women who are pregnant and/or lactating. 2) Significant Medical History: History or presence of significant cardiovascular (including QT prolongation, clinically significant hypokalemia, or other proarrhythmic conditions), pulmonary, hepatic, renal, hematological, gastrointestinal, endocrine (including glucose intolerance, diabetes mellitus), immunologic (including asthma or seasonal allergies [that require intermittent use of steroids or other medication]), musculoskeletal (including tendinopathy), dermatologic, or neurological disease (including seizure disorders, psychiatric disorders), including any acute illness or surgery within the past 3 months, as determined by the Investigator to be clinically relevant.

     1. History of any kidney disease or current or chronic history of impaired renal function as indicated by a calculated creatinine clearance (Cockcroft-Gault formula) <80 milliliter per minute (mL/min).
     2. Current or chronic history of liver disease or known hepatic or biliary abnormalities (except for Gilbert syndrome or asymptomatic gallstones) 3) Laboratory abnormalities

     a) Clinically significant abnormal findings in serum chemistry, hematology, coagulation or urinalysis results obtained at screening or check-in (Day-1) b) Alanine aminotransferase (ALT) more than (>)1 upper limit of normal (ULN) at screening or check-in (Day-1) c) Aspartate aminotransferase (AST) > ULN at screening or check-in (Day-1)d) Bilirubin >ULN at screening or check-in (Day-1) e) Serum creatinine > ULN at screening or check-in (Day-1). The serum creatinine or any laboratory test may be repeated prior to confirming exclusion, at the PI's discretion.

     4) Electrocardiographic abnormalities: Baseline QTcF of >450 msec (for males), and >470 msec (for females) at screening or check-in (Day-1) 5) Photosensitivity: History of photosensitivity to quinolones 6) Clostridium Difficile: History of known or suspected Clostridium difficile infection 7) Hospitalization History: Any condition that necessitated hospitalization within the 3 months prior to Day -1 or is likely to require so during the study 8) Antibiotic History: No systemic antibiotic use within 5 days before dosing. 9) Infection History: Positive test for hepatitis B virus surface antigen (HBsAg), hepatitis C virus antibody (anti-HCV antibodies), or human immunodeficiency virus antibody (antibodies to HIV-1, HIV-2) at screening.

     10) Recent Medications: Exclude participants receiving all prescription and OTC medications (except hormonal contraception and Paracetamol) 14 days or 5 half-lives, whichever is longer, prior to IP dosing.Discussion between the PI and the Sponsor Medical Monitor is encouraged regarding prior use of any medications during the pre-dose period. Note: An exception is made for hormonal contraceptives, paracetamol (a maximum of 4 doses per day of 500 mg, and no more than 3 g per week) for the treatment of headache or any other pain as per the PI's judgement.

     11) Hypersensitivity: DocumentedHistory of significant hypersensitivity reaction or anaphylaxis to any medication, as determined by the Medical Officer.

     12) Tobacco and Nicotine Use: Smoker (including tobacco, e-cigarettes, or marijuana) or nicotine user within 1 month prior to dosing and have a positive test for cotinine at check in on Day -1 (may be repeated once, at the discretion of the Investigator or Medical officer, in the instance of a positive result).

     13) Drug/Alcohol Abuse: Positive urine drug/alcohol breath testing at screening or check-in (Day -1), or history of substance abuse or alcohol abuse (defined as greater than 2 standard drinks on average each and every day, where one standard drink is defined as containing 10 g of alcohol and is equivalent to 1 can or stubby of mid-strength beer, 30 ml nip spirits, or 100 ml wine) within the previous 5 years (may be repeated once per timepoint, at the discretion of the Investigator or Medical officer, in the instance of a positive result).

     14) Blood/Plasma Donation: Donation of blood within 30 days or plasma within 7 days prior to randomization, or loss of whole blood of more than 500 mL within 30 days prior to randomization, or receipt of a blood transfusion within 1 year of study enrollment.

     15) Previous Study Participation: Previous participation in this study, i.e., who has already completed earlier cohorts or previous participation in another study within 5 half-lives (if known) of the agent, or 30 days, whichever is longer, of Day 1.

   Note: prior participation at any time in non-invasive methodology trials in which no drugs were given is acceptable. Those who were screen failures or not dosed in this study may will be considered for re-screening in subsequent cohorts.

16) Food Restrictions: Consumption of red wine, Seville oranges, grapefruit, or grapefruit juice, pummelos, exotic citrus fruits, grapefruit hybrids, or fruit juices containing such products from 7 days prior to the first dose of study medication.(Note: Lemon and lime, including their juice or zest, are permitted as they are not known to significantly affect cytochrome P450 (CYP3A4) enzyme activity) 17) Sponsor Relationships: Employee or family member of an employee of the Sponsor, CRU, or clinical research organization at which the study will be conducted.

18) Non-compliance: Unable to cooperate fully with the requirements of the study protocol, including the schedule of events, or likely to be non-compliant with any study requirements.

19) Other Medical Conditions: Any other disease or condition that, in the opinion of the Investigator, would preclude the subject's participation in the study or place them at risk as a result of study participation.

Note: Volunteers should refrain from consumption of any foods containing poppy seeds within 48 hours (2 days) prior to screening and prior to Day -1 to avoid false positive drug screen results. Examples of foods to avoid include: poppy seed bagels, muffins, pastries, salad dressings, or any baked goods or dishes that list poppy seeds as an ingredient.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Estimated)
Dates: Start 2025-10-10 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-08-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of treatment-emergent adverse events (TEAEs and serious adverse events (SAEs) overall and by intensity (Safety and tolerability). | SAD: Up to 8 days MAD: Up to 16 days
  Description: This outcome combines the measure of the number of participants experiencing adverse events (AEs), the nature and severity of those AEs and their relationship to the study treatment.

SECONDARY OUTCOMES:
AUC[0-t] of BWC0977 following single dose administration | Immediately before (within 60 minutes before) the start of infusion of the study drug and 5, 10,15, 20, 30, 45, 60, 75, and 90 minutes, 2, 2.5, 3, 4, 6, 8, 10, 12, 24 and 48 hours after the start of study drug infusion.
  Area under the plasma concentration curve from time zero to last time of quantifiable concentration (AUC0-t) of BWC0977 following single dose administration
AUC[0-inf] of BWC0977 following single dose administration | Immediately before (within 60 minutes before) the start of infusion of the study drug and 5, 10,15, 20, 30, 45, 60, 75, and 90 minutes, 2, 2.5, 3, 4, 6, 8, 10, 12, 24 and 48 hours after the start of study drug infusion.
  Area under the plasma concentration curve from time zero to infinity (AUC0-inf) of BWC0977 following single dose administration
AUC[0-8], AUC[0-12], AUC[0-24] of BWC0977 following single dose administration | Immediately before (within 60 minutes before) the start of infusion of the study drug and 5, 10,15, 20, 30, 45, 60, 75, and 90 minutes, 2, 2.5, 3, 4, 6, 8, 10, 12, 24 and 48 hours after the start of study drug infusion.
  AUC from time zero to 8, 12, and 24 hours (AUC[0-8], AUC[0-12], AUC[0-24]) of BWC0977 following single dose administration
Cmax of BWC0977 following single dose administration | Immediately before (within 60 minutes before) the start of infusion of the study drug and 5, 10,15, 20, 30, 45, 60, 75, and 90 minutes, 2, 2.5, 3, 4, 6, 8, 10, 12, 24 and 48 hours after the start of study drug infusion.
  Maximum observed plasma concentration (Cmax) of BWC0977 following single dose administration
Cmax of BWC0977 following repeated dose administration | Immediately before (within 60 minutes before) the start of the first infusion and at 5,15, 30, 60, 75, and 90 minutes, 2, 4, 6, and 8, 12, 24 hours after the start of the last infusion on Day 1 and 7 (MAD 1 cohort) or 10 (For MAD2 -MAD4 cohort).
  Maximum observed plasma concentration (Cmax) of BWC0977 following repeat dose administration
Termianl Half life (T1/2) of BWC0977 following single dose administration | Immediately before (within 60 minutes before) the start of infusion of the study drug and 5, 10,15, 20, 30, 45, 60, 75, and 90 minutes, 2, 2.5, 3, 4, 6, 8, 10, 12, 24 and 48 hours after the start of study drug infusion.
  Terminal half-life (T1/2) of BWC0977 following single dose administration
Systemic clearance (CL) following single dose administration | Immediately before (within 60 minutes before) the start of infusion of the study drug and 5, 10,15, 20, 30, 45, 60, 75, and 90 minutes, 2, 2.5, 3, 4, 6, 8, 10, 12, 24 and 48 hours after the start of study drug infusion.
  Systemic clearance (CL) of BWC0977 following single dose administration
Volume of distribution at steady state (Vdss) following single dose administration | Immediately before (within 60 minutes before) the start of infusion of the study drug and 5, 10,15, 20, 30, 45, 60, 75, and 90 minutes, 2, 2.5, 3, 4, 6, 8, 10, 12, 24 and 48 hours after the start of study drug infusion.
  Volume of distribution at steady state (Vdss) of BWC0977 following single dose
Pre-dose (trough) concentration (Ct) at the end of the dosing interval | Immediately before (within 60 minutes before) the start of the first infusion and at 5,15, 30, 60, 75, and 90 minutes, 2, 4, 6, and 8, 12, 24 hours after the start of the last infusion on Day 1 and 7 (MAD 1 cohort) or 10 (For MAD2 -MAD4 cohort).
  Pre-dose (trough) concentration (Ct) at the end of the dosing interval of BWC0977 following repeat dose administration
Volume of distribution at steady state following repeat dose administration | Immediately before (within 60 minutes before) the start of the first infusion and at 5,15, 30, 60, 75, and 90 minutes, 2, 4, 6, and 8, 12, 24 hours after the start of the last infusion on Day 1 and 7 (MAD 1 cohort) or 10 (For MAD2 -MAD4 cohort).
  Volume of distribution at steady state (Vdss) of BWC0977 following repeat dose
Observed accumulation ratio following repeat dose administration | Immediately before (within 60 minutes before) the start of the first infusion and at 5,15, 30, 60, 75, and 90 minutes, 2, 4, 6, and 8, 12, 24 hours after the start of the last infusion on Day 1 and 7 (MAD 1 cohort) or 10 (For MAD2 -MAD4 cohort).
  Observed accumulation ratio (Ro) of BWC0977 following repeat dose administration
Amount excreted in urine (Ae) following repeat dose administration | Day 1 pre-dose, 0-8 hours post infusion start Day 7 (MAD1 Cohort): 0-12 hours post infusion start Day 10 (MAD 2-3 cohort): 0-12 hours post infusion start Day 10 (MAD 4 Cohort): 0-8 hours post infusion start
  Amount excreted in urine (Ae) of BWC0977 following repeat dose administration
Amount excreted in urine (Ae) following single dose administration | 0-4, 4-8, >8-12, >12-24 hours (Days 1-2), >24-36, and >36-48 hours (Days 2-3) after the start of the study drug infusion.
  Amount excreted in urine (Ae) of BWC0977 following single dose administration
Fraction of the dose excreted in urine (fe) following single dose administration | 0-4, 4-8, >8-12, >12-24 hours (Days 1-2), >24-36, and >36-48 hours (Days 2-3) after the start of the study drug infusion.
  Fraction of the dose excreted in urine (fe) of BWC0977 following single dose administration
Fraction of the dose excreted in urine (fe) following repeat dose administration | Day 1 pre-dose, 0-8 hours post infusion start Day 7 (MAD1 Cohort): 0-12 hours post infusion start Day 10 (MAD 2-3 cohort): 0-12 hours post infusion start Day 10 (MAD 4 Cohort): 0-8 hours post infusion start
  Fraction of the dose excreted in urine (fe) of BWC0977 following repeat dose administration
Renal Clearance (CLr) following single dose administration | 0-4, 4-8, >8-12, >12-24 hours (Days 1-2), >24-36, and >36-48 hours (Days 2-3) after the start of the study drug infusion.
  Renal Clearance (CLr) of BWC0977 following single dose administration
Renal Clearance (CLr) following repeat dose administration | Day 1 pre-dose, 0-8 hours post infusion start Day 7 (MAD1 Cohort): 0-12 hours post infusion start Day 10 (MAD 2-3 cohort): 0-12 hours post infusion start Day 10 (MAD 4 Cohort): 0-8 hours post infusion start
  Renal Clearance (CLr) of BWC0977 following repeat dose administration

CONTACTS AND LOCATIONS:
Locations (1):
- Nucleus Network, Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: Undecided